CLINICAL TRIAL: NCT01226355
Title: Clinical Trial Program of a Medical Instrument Product
Brief Title: NOYA CoCr Biodegradable Coating Sirolimus-Eluting Coronary Stent System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medfavour (Beijing) Medical Co., Ltd (Industry)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Division of Biometrics,National Center for Cardiovascular Diseases,China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FW2009-183
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Diseases
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOYA (Experimental): implant NOYA CoCr Biodegradable Coating Sirolimus-Eluting Stents Intervention: Device: stent
  Interventions: Device: stent
- Firebird2 (Active Comparator): implant Firebird2 drug-eluting stents Intervention: Device: stent
  Interventions: Device: stent

INTERVENTIONS:
Device: stent — NOYA CoCr Biodegradable Coating Sirolimus-Eluting Stent System is manufactured by Medfavour (Beijing) Medical Co., Ltd.
  Firebird drug-eluting stents from MicroPort Medical (Shanghai) Co., Ltd.
  Other Names: NOYA CoCr Biodegradable Coating Sirolimus-Eluting Stent System; Firebird2 drug-eluting stents

SUMMARY:
A single blind, multi-center, randomized study is preformed to compare NOYA CoCr biodegradable coating sirolimus-eluting stents with Firebird2 drug-eluting stents from MicroPort Medical (Shanghai) Co., Ltd. to evaluate the safety and efficacy of NOYA CoCr biodegradable coating sirolimus-eluting stents in treating coronary artery lesions.

DETAILED DESCRIPTION:
A single blind, multi-center, randomized study is preformed to compare NOYA CoCr biodegradable coating sirolimus-eluting stents with Firebird2 drug-eluting stents from MicroPort Medical (Shanghai) Co., Ltd. to evaluate the safety and efficacy of NOYA CoCr biodegradable coating sirolimus-eluting stents in treating coronary artery lesions. Appropriate patients judged by inclusion and exclusion standards will be preformed stent implantation, and after that all patients will be clinically followed up at 30, 90, 180, 270,365 days,2 years,3 years,4 years and 5 years. Especially, standard quantity coronary angiography (QCA) will be conducted at 270 days (±30days) through which the main therapeutic indicator of late luminal loss (LLL) is obtained so as to evaluate the efficacy of tested stents. Major adverse cardiac events (MACEs) found in following-up period as key indicators to evaluate the safety of stents. The arrangement, conclusion and statistical analysis of trial data including clinography and angiography will be fulfilled by independent Data Management Center(DMC) and radiography core laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, men or unpregnant women;
2. Angina pectoris patients with non-symptom myocardial ischemia, or patients with obsolete myocardial infarction;
3. Total of lesion artery ≤2;
4. Lesion artery ≤30 mm in length, 2.25 to 4.0 mm in diameter (ocular estimate);
5. Narrow level of lesion artery ≥70% in diameter (ocular estimate);
6. Amount of same stents implanted in a lesion artery ≤2;
7. Patients with indications of coronary artery bridging surgery(coronary artery bypass transplant technique);
8. Patients knowing about the objective of trial, willing to sign a statement of informed consent and join in this trial, and willing to accept follow-up.

Exclusion Criteria:

1. Patients with acute myocardial infarction in 7 days;
2. Chronic total occlusion lesions(TIMI 0 grade blood flow prior to implantation), left trunk vessel lesion, three-branch lesions needing treated, fork and bridge vessel lesions of branch vessels whose diameter ≥2.25mm;
3. Severe calcific lesions and twisted lesions which cannot be pre-expanded, and lesions unsuitable for delivering and expanding stents;
4. In-stent restenosis lesions;
5. Patients with stent implantation in his/her coronary artery within recent one year;
6. Severs heart failure(over NYHA III grade ), or left ventricular ejection fraction(LVEF)< 40%( supersonic inspection or left ventricular radiography );
7. Kidney functional damage prior to implantation, serum creatinine level>2.0mg/dl;
8. Patients with hemorrhage tendency, an active digestive ulcer history, a cerebral hemorrhage or subarachnoid hemorrhage history, or cerebral apoplexy within half a year, and these patients who contraindicate against platelet inhibitors and anticoagulant therefore can not bear anticoagulation treatment;
9. Patients allergic to aspirin, clopidogrel or ticlopidine, heparin, contrast medium, rapamycin and metals;
10. Patients whose life expectancy less than 12 months;
11. Patients who are participating in other drugs or medical devices clinical trials;
12. Patients who can not comply with the clinical trial protocol;
13. Patients having a heart transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
In-stent late loss at 9-month | 270 days (±30days)
  Standard quantity coronary angiography (QCA) will be conducted at 270 days (±30days) through which the main therapeutic indicator of late luminal loss (LLL) is obtained so as to evaluate the efficacy of tested stents.

SECONDARY OUTCOMES:
MACEs found in follow-up period | 5 years
  Major adverse cardiac events (MACEs) found in following-up period as key indicators to evaluate the safety of stents.

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Professor, Principal Investigator — Fu Wai Hospital, National Center for Cardiovascular Diseases,China
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Beijing, China

REFERENCES:
- [Derived] Xu B, Dou K, Yang Y, Lv S, Wang L, Wang H, Li Z, Wang L, Chen Y, Huo Y, Li W, Kirtane AJ, Gao R. Nine-month angiographic and 2-year clinical follow-up of the NOYA biodegradable polymer sirolimus-eluting stent in the treatment of patients with de novo native coronary artery lesions: the NOYA I trial. EuroIntervention. 2012 Nov 22;8(7):796-802. doi: 10.4244/EIJV8I7A122. PMID 23171800